CLINICAL TRIAL: NCT02677987
Title: Treating Cognitive Impairments in Cancer Patients Via Systematic Light Exposure
Brief Title: The "Light for the Brain" Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisa M. Wu, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00201700; 7K07CA184145-02 (NIH)
Record Dates: First submitted 2016-01-22; First posted 2016-02-09 (Estimated); Results first posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-03

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cognitive Impairments; Sleep; Depression; Fatigue; Quality of Life
MeSH Terms: conditions — Cognitive Dysfunction; Depression; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention light (Experimental): 30 minutes of intervention systematic light exposure daily for 4 weeks.
  Interventions: Device: Intervention systematic light exposure
- Comparison light (Active Comparator): 30 minutes of comparison systematic light exposure daily for 4 weeks.
  Interventions: Device: Comparison systematic light exposure

INTERVENTIONS:
Device: Intervention systematic light exposure — Bright light using Litebook device.
  Arms: Intervention light
Device: Comparison systematic light exposure — Dim light using modified Litebook device.
  Arms: Comparison light

SUMMARY:
Cognitive impairment (such as memory problems) due to cancer and its treatment can interfere with quality of life and can linger long after treatment has ended, yet research examining cognitive rehabilitation approaches has produced limited clinical benefit. The proposed study will provide information about systematic light exposure for the treatment of cognitive impairment in hematopoietic stem cell transplant (HSCT) survivors and will investigate how it works. This study would facilitate the development of this potential treatment, giving health care providers and cancer survivors a much-needed tool to help with cancer-related cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Have a history of HSCT,
2. 1 to 5 years post-HSCT,
3. Relapse-free since most recent HSCT,
4. Age 21 or older,
5. English language proficient
6. Able to provide informed consent
7. Endorse subjective cognitive impairment.

Exclusion Criteria:

1. Diagnosed or suspected neurological, psychiatric (including bipolar disorder or mania), or medical condition that might impair cognitive functioning (other than those caused by the cancer or its treatment),
2. Visual, hearing, or physical impairment sufficient to interfere with cognitive testing or participation,
3. Have a history of whole brain irradiation or surgery,
4. Active diagnosis of autoimmune and/or inflammatory disorder or disorders that may influence immune processes,
5. Chronic use of oral steroid medication,
6. History of systematic light exposure treatment,
7. Diagnosed sleep apnea or narcolepsy,
8. Use of photosensitizing medications,
9. Plan to travel across meridians during the study,
10. Work night, early morning, or swing shifts,
11. Adults unable to consent, individuals who are not yet adults, pregnant women and prisoners will be excluded from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Wu, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu LM, Valdimarsdottir HB, Amidi A, Reid KJ, Ancoli-Israel S, Bovbjerg K, Fox RS, Walker L, Matharu A, Kaseda ET, Galvin JP, Adekola K, Winkel G, Penedo F, Redd WH. Examining the Efficacy of Bright Light Therapy on Cognitive Function in Hematopoietic Stem Cell Transplant Survivors. J Biol Rhythms. 2022 Oct;37(5):471-483. doi: 10.1177/07487304221107833. Epub 2022 Jul 29. PMID 35904252

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparison Light: 30 minutes of comparison long wavelength systematic light exposure daily for 4 weeks.
  Comparison systematic light exposure: Dim light using modified Litebook device.
Period: Overall Study
Arm/Group | Intervention Light | Comparison Light
Started | 23 | 24
Completed | 19 | 24
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Light | Comparison Light | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.2) | 55.5 (13.0) | 56.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 6 | 11 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 21 | 23 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47
Wechsler Test of Adult Reading [Mean (Standard Deviation); unit: units on a scale] — Baseline estimate of premorbid intellectual functioning; The WTAR (Wechsler, 2001) comprises 50 words with irregular pronunciations that participants read aloud. The raw score ranges from 0 to 50, with a higher score indicating better performance, and the raw score can be transformed to an age-adjusted standard score, which is used to predict IQ (M = 100; SD = 15).
  units on a scale | 105.6 (9.5) | 110.3 (11.1) | 108.0 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Functioning (Neuropsychological Tests)
Description: Global composite z-score from baseline to 8 weeks after the intervention based on the HVLT-R; BVMT-R; Psychomotor vigilance task; Trail-making tests A and B; WAIS-IV Coding, Digit Span, Block Design; D-KEFS Color-Word Inhibition, Verbal Fluency; Conners Continuous Performance Test III.
  Raw scores at baseline of tests within single domains were averaged and then standardized to z-scores. The mean of the z-scores was calculated, and then this composite z-score was standardized to z-scores. Follow up intervention z-scores were calculated based on differences between raw scores at baseline and raw scores at follow-up time points and divided by the standard deviation of the baseline domain z-score) within each domain, and then averaged to create follow up global composite scores.
  A z-score below 0 indicated poorer performance than at baseline and a z-score above 0 indicated better performance than at baseline.
Time Frame: Baseline to end-of-intervention to 8 weeks after the intervention
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Intervention Light | Comparison Light
Number analyzed (Participants) | 21 | 18
z-score
  End of intervention | 0.24 (0.14) | 0.16 (0.14)
  8 weeks after intervention | 0.43 (0.14) | 0.50 (0.14)

2. Secondary Outcome: Circadian Activity Rhythms (Actigraphy)
Description: F statistic from actigraphy was assessed as a measure of circadian activity rhythm robustness.
Time Frame: Baseline to end of intervention to 8 weeks later
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Light | Comparison Light
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline | 1696.19 (290.49) | 1551.72 (293.04)
  End of intervention | 1999.72 (295.87) | 1373.88 (293.04)
  8 weeks after intervention | 1858.04 (293.04) | 1466.82 (295.87)

3. Secondary Outcome: Sleep Quality (Pittsburgh Sleep Quality Index)
Description: The Pittsburgh Sleep Quality Index consists of 19 self-rated items used to calculate sleep quality
Time Frame: Baseline, mid intervention, end of intervention, 8 weeks later
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 24 | 20
units on a scale
  Baseline | 7.3157 (0.7672) | 8.5000 (0.6910)
  Mid-treatment | 6.7500 (0.8544) | 7.7500 (0.7137)
  End of treatment | 6.5296 (0.7567) | 7.5500 (0.6343)
  8 weeks later | 6.1922 (0.7345) | 8.3745 (0.8023)

4. Secondary Outcome: Fatigue (FACIT-fatigue)
Description: This is a 13-item measure of fatigue.
Time Frame: Baseline, mid-intervention, end of the intervention, 8 weeks later
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 24 | 20
units on a scale
  Baseline | 29.9804 (1.7374) | 30.0000 (1.5458)
  Mid-intervention | 29.5833 (2.1666) | 33.6356 (1.3701)
  End of intervention | 30.8219 (1.9725) | 33.7513 (1.4237)
  8 weeks post-intervention | 30.5041 (2.1484) | 32.3366 (1.8079)

5. Secondary Outcome: Depressed Mood (CESD)
Description: The Center for Epidemiological Studies Depression Scale (CES-D) is a 20-item self-report instrument that measures symptoms of depressed mood over the past week.
Time Frame: Baseline, Mid-intervention, End of intervention, 8 weeks later
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 24 | 23
units on a scale
  Baseline | 18.6293 (1.3655) | 20.4500 (1.4378)
  Mid-intervention | 20.4583 (1.5343) | 18.1000 (1.0366)
  End of intervention | 19.1489 (1.2097) | 17.0500 (1.1821)
  8 weeks post intervention | 20.1206 (1.6286) | 19.0299 (1.1423)

6. Secondary Outcome: Neurobehavioral Functioning (Frontal Systems Behavioral Scale)
Description: Total raw score for entire scale (minimum = 46, maximum = 230) with a higher score indicating greater neurobehavioral symptomatology.
Time Frame: Baseline, mid-intervention, end-of-intervention, 8 weeks later
Population: Participants did not always complete this measure, which accounts for why there are sometimes fewer participants than the overall number of participants analyzed at different time points. Linear mixed models allows for missing time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 24 | 22
score on a scale
  Baseline: number analyzed (Participants) | 23 | 22
  Baseline | 91.39 (17.71) | 89.36 (19.57)
  Mid-intervention: number analyzed (Participants) | 24 | 20
  Mid-intervention | 92.96 (21.12) | 90.55 (18.56)
  End-of-intervention: number analyzed (Participants) | 23 | 20
  End-of-intervention | 89.04 (19.69) | 88.90 (19.08)
  8 weeks later: number analyzed (Participants) | 24 | 18
  8 weeks later | 87.29 (21.58) | 92.78 (19.47)

7. Secondary Outcome: Quality of Life (FACT-BMT)
Description: This 50-item scale is a commonly used and well-validated measure of the functional status of cancer patients who have undergone BMT (SCT).
Time Frame: Baseline, End of intervention, 8 weeks post-intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Light | Comparison Light
Number analyzed (Participants) | 23 | 20
units on a scale
  Baseline | 110.27 (4.1870) | 109.66 (4.2157)
  End of intervention | 116.88 (3.5606) | 111.94 (4.9821)
  8 weeks post-intervention | 112.68 (4.4154) | 110.92 (5.0970)

8. Secondary Outcome: Interleukin-6
Description: Serum cytokine IL-6 in pg/mL
Time Frame: Baseline and end-of-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 23 | 18
units on a scale
  Baseline | 3.24 (2.72) | 3.24 (1.79)
  End-of-intervention | 3.98 (4.87) | 3.28 (2.60)

9. Secondary Outcome: Pro-inflammatory Cytokine - TNF Alpha
Description: Serum cytokine TNF-α in pg/mL
Time Frame: Baseline and end-of-intervention
Population: Two participants did not provide blood samples at the end-of-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 23 | 18
units on a scale
  Baseline | 7.55 (2.49) | 7.00 (2.13)
  End-of-intervention: number analyzed (Participants) | 21 | 18
  End-of-intervention | 7.44 (3.26) | 7.30 (2.36)

10. Secondary Outcome: C-Reactive Protein
Description: C-reactive protein in mg/L
Time Frame: Baseline and end-of-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 23 | 18
units on a scale
  Baseline | 5.67 (10.11) | 3.68 (3.09)
  End-of-intervention | 5.95 (15.29) | 3.53 (2.61)

11. Secondary Outcome: Self-reported Cognitive Function (Patient Assessment of Own Functioning Inventory)
Description: The 33-item Patient Assessment of Own Functioning Inventory (PAOFI) is a reliable and valid measure of perceptions of cognitive functioning (Bell et al., 2013; Chelune et al., 1986). Using a Likert scale from 1 (Almost Always) to 6 (Almost Never), ratings of 1-3 were scored "1" indicating impairment, and ratings from 4 to 6 were scored "0" indicating no impairment. Total impairment was calculated by summing the number of impaired items.
Time Frame: Baseline, mid-intervention, end of intervention, 8 weeks after intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Light | Comparison Light
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline | 8.5217 (1.219) | 7.9703 (1.2023)
  Mid-intervention | 6.5927 (1.2457) | 6.9583 (1.1934)
  End of intervention | 4.7065 (1.258) | 5.5905 (1.2023)
  8 weeks after intervention | 7.0445 (1.284) | 6.2142 (1.2023)

12. Other Pre Specified Outcome: Treatment Satisfaction (FACT-TS)
Description: Range between 0 and 5, with 5 meaning higher treatment satisfaction
Time Frame: During the 4th week of the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Light | Comparison Light
Number analyzed (Participants) | 23 | 24
units on a scale | 2.5 (0.8) | 2.0 (1.0)

13. Other Pre Specified Outcome: Credibility/Expectancy (Credibility/Expectancy Questionnaire)
Description: Treatment credibility and outcome expectancy were assessed at baseline with the mean of the first 3 items of the Credibility/Expectancy Questionnaire. Items are scored on a Likert scale from 1 to 9, and the term "symptoms" was replaced with "thinking, memory and concentration problems." Higher scores represent greater credibility and outcome expectancy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 24 | 23
units on a scale | 6.9 (1.5) | 6.3 (1.4)

14. Other Pre Specified Outcome: Usage of Light Box (Integrated Meter Measurement and Litebook Log)
Description: Length of time light box has been used.
Time Frame: Throughout intervention period (4 weeks)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 24 | 23
days | 21.1 (7.5) | 21.0 (8.7)

15. Other Pre Specified Outcome: Chronotype (Morningness-eveningness Questionnaire)
Description: Measure determines chronotype with a lower score indicating an evening type and a higher score indicating a morning type.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comparison Light | Intervention Light
Number analyzed (Participants) | 23 | 20
score on a scale | 17.91 (3.15) | 15.65 (4.11)

ADVERSE EVENTS:
Time Frame: 13 to 16 weeks
Arm/Group | Intervention Light | Comparison Light
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT02677987/Prot_SAP_ICF_000.pdf